CLINICAL TRIAL: NCT04822805
Title: Anlotinib in the Treatment of Recurrent High-grade Glioma： an Open-label Single-arm, Phase 2 Trials
Brief Title: A Study of Anlotinib in the Treatment of Recurrent High-grade Glioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2CH2020M504
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Recurrent High-grade Glioma
MeSH Terms: conditions — Glioma | interventions — anlotinib

STUDY DESIGN:
Intervention Model Description: Patients with recurrent high-grade gliomas are being enrolled , treated with anlotinib , and being observed the disease-related outcomes of the patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with Anlotinib (Experimental): Patients with recurrent high-grade gliomas are being enrolled , treated with anlotinib 12mg once daily for 14 days every 3 weeks until disease progression or unacceptable toxicity.The dose can be adjusted to 10mg or 8mg according to the specific conditions of the patient.
  Interventions: Drug: Anlotinib hydrochloride

INTERVENTIONS:
Drug: Anlotinib hydrochloride — Patients with recurrent high-grade gliomas are being enrolled , treated with anlotinib 12mg once daily for 14 days every 3 weeks until disease progression or unacceptable toxicity.The dose can be adjusted to 10mg or 8mg according to the specific conditions of the patient.
  Other Names: Anlotinib

SUMMARY:
This is a phase II, open-label, single center study, aiming to investigate safety and efficacy of anlotinib in treatment of recurrent high-grade glioma.

DETAILED DESCRIPTION:
Glioma is a common primary central nervous system malignant tumor that originates from glial cells. High grade glioma (HGG) refers to grade III and IV gliomas in the central nervous system tumor classification of the World Health Organization (WHO), accounting for approximately 67% of newly diagnosed cases. The maximum safety resection of the tumor followed by radiotherapy and chemotherapy is the HGG standard initial treatment strategy. However, glioma cells grow aggressively, and most patients will relapse after initial treatment. Recurrent high-grade glioma (r-HGG) is difficult to treat, lacking treatment standards and having a poor prognosis.

There is no standard treatment plan for patients with recurrent high-grade cancer. Studies have shown that gliomas highly express a variety of pro-angiogenic factors and have a large number of abnormally proliferated blood vessels, VEGF especially playing an important role in the formation of GBM neovascularization. VEGF is almost not expressed in normal tissues, but it is highly expressed (about 96%) in malignant gliomas and surrounding tissues, especially VEGF-A is highly expressed in glioblastomas. Therefore, VEGF It can be used as an effective target for anti-angiogenesis treatment of malignant glioma.

Anlotinib hydrochloride is a multi-target receptor tyrosine kinase inhibitor that has significant inhibitory activity against angiogenesis related kinases such as VEGFR1/2/3, FGFR1/2/3, and other tumor related kinases such as PDGFR /, C-Kit, Ret, etc. (e.g., Met, FGFR1/2/3).

Based on the above theory , the purpose of this study was to explore the efficacy and safety of anlotinib in treatment of recurrent high-grade glioma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old (calculated on the day of signing the informed consent), regardless of gender.
2. Karnofsky score (KPS score) ≥60.
3. According to Rano criteria, there are evaluable intracranial lesions, and recurrent high-grade gliomas have been confirmed.
4. Patients have undergone surgery and relapsed after receiving standard radiotherapy and chemotherapy;
5. The toxicity has returned to ≤1 grade If have received chemotherapy;
6. Expected survival ≥ 3 months;
7. The patient has no major organ dysfunction. Specific laboratory indicators are required: white blood cells ≥3.0×109/L, platelets ≥75×109/L, hemoglobin ≥10g/dl, and serum bilirubin not greater than 1.5 times the maximum normal value; ALT and AST are not more than 2 times the maximum normal value; blood creatinine ≤ 1.5 mg/dl.
8. Men and women of gestational age must agree to take adequate contraceptive measures throughout the study period.
9. The patient voluntarily joined the study and signed a written informed consent.

Exclusion Criteria:

1. Those who have multiple factors that affect oral medications (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
2. Patients with any severe and/or uncontrollable disease, including:

1) Patients with unsatisfactory blood pressure control (systolic blood pressure ≥150 mmHg, diastolic blood pressure ≥100 mmHg); 2) Patients with myocardial ischemia or myocardial infarction above grade I, arrhythmia (including QTC ≥480ms), and grade ≥2 congestive heart failure (New York Heart Association (NYHA) classification); 3) Active or uncontrolled serious infection (≥CTC AE Grade 2 infection); 4) Liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral treatment; 5) Renal failure requires hemodialysis or peritoneal dialysis; 6) Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; 7) Diabetes is poorly controlled (fasting blood glucose (FBG)> 10mmol/L); 8) Urine routines suggest that urine protein is ≥++, and the 24-hour urine protein quantification is more than 1.0 g; 9) Patients who have seizures and need treatment; 3. Received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before enrollment; 4. Patients whose imaging shows that the tumor has invaded important blood vessels or the researcher judges that the tumor is likely to invade important blood vessels causing fatal hemorrhage during the follow-up study; 5. Regardless of the severity, patients with any signs of bleeding or medical history; within 4 weeks before enrollment, patients with any bleeding or bleeding event ≥ CTCAE level 3, unhealed wounds, ulcers or fractures; 6. Those who have had arterial/venous thrombosis within 6 months, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis and pulmonary embolism; 7. Those who have a history of psychotropic drug abuse and cannot be quit or have mental disorders; 8. Participated in clinical research of other anti-tumor drugs within four weeks; 9. Have received the treatment of small molecule anti-angiogenesis targeted drugs (such as regorafenib, perzopanib, apatinib, etc.); 10. Those considered by the researcher to be unsuitable for inclusion。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 5months
  The time interval from the randomization of the patient to the first disease progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Hui Dai, Principal Investigator — Hangzhou Cancer Hospital
Locations (1):
- Hangzhou Cancer Hospital, Hangzhou, China

REFERENCES:
- [Derived] Zhao S, Zhang M, Zhang Q, Wu J, Dai H. Anlotinib alone or in combination with bevacizumab in the treatment of recurrent high-grade glioma: a prospective single-arm, open-label phase II trial. BMC Cancer. 2024 Jan 2;24(1):6. doi: 10.1186/s12885-023-11776-4. PMID 38166698